CLINICAL TRIAL: NCT06713863
Title: Intervention Effectiveness Study of BEtter AT LEarning (BEATLE)- Digital Neuropsychological Rehabilitation Program
Acronym: BEATLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Sari-Anne Levänen, PhD, Neuropsychologist, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HUS/6774/2023
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Dyslexia, Developmental; Developmental Language Disorder; Specific Learning Disorder; Borderline Intellectual Functioning
Keywords: eHealth; Adolescence; Intervention; Effectiveness; RCT
MeSH Terms: conditions — Dyslexia; Language Development Disorders; Specific Learning Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention first (Experimental): Participant directly enrolled to the intervention
  Interventions: Other: BEtter AT LEarning (BEATLE)- Digital Care Pathway
- Waitlist first (No Intervention): Participant spends amount of time similar to completing the intervention in a waitlist after which gets enrolled into the intervention after post-waitlist measures have been completed.

INTERVENTIONS:
Other: BEtter AT LEarning (BEATLE)- Digital Care Pathway — BEATLE is a digital care pathway consisting of ten episodes resembling an online course. The episodes are designed to be multimodal and immersive, incorporating text, recorded voice, pictures, cartoons, videos and peer support through given examples and case stories. Participants are encouraged to access BEATLE through a web browser on a computer, although it is also accessible through a mobile application. Participants have control over the pace of completing the BEATLE, but there must be a minimum five-day break between episodes. In other words, it is possible to complete the BEATLE in seven weeks.
  All participants are referred to the BEATLE by a neuropsychologist and are strongly authenticated in the healthvillage.fi online platform. Each participant is assigned a designated neuropsychologist who tracks their progress in the BEATLE and to whom messages and questions can be sent by the participant.
  Arms: Intervention first

SUMMARY:
The purpose of this study is to evaluate the effectiveness of BEATLE with clinical samples of patients diagnosed with Developmental Language Disorder (DLD), Dyslexia, and Mixed Specific Developmental Disorder. A randomized controlled trial with a waitlist design will be employed. The objective is to assess potential changes in perceived self-efficacy, self-compassion, executive functioning, and attitudes toward learning as reported by the participants, their guardians (parents), and teachers. Additionally, this study aims to examine the correlation between the usage of the Digital Care Pathway (DCP) and its effectiveness.

DETAILED DESCRIPTION:
BEATLE (BEtter AT LEarning) is a neuropsychological digital rehabilitative program (Digital Care Pathway, DCP) developed at the Department of Phoniatrics, University Hospital of Helsinki and Uusimaa region (HUS). The purpose of this DCP is to provide knowledge on meta-skills and tools for learning to 12-16-year-olds who experience learning difficulties due to developmental language disorder, dyslexia, or other developmental issues.

The aforementioned developmental disorders can have long-lasting impacts on individuals' lives. For instance, children with DLD have been reported to have a lower quality of life than typically developing children, according to parent evaluations. Self-evaluation is a crucial aspect of individual performance and well-being. Albert Bandura's social cognitive theory posits that individuals are proactive and reflective beings who simultaneously shape and are shaped by their environment (Reciprocal Determinism). According to Bandura, individuals constantly evaluate and form beliefs about their capabilities to perform in given situations (Self-efficacy). The theory of self-efficacy is often employed in educational sciences, where students with higher self-efficacy beliefs have been found to exert more effort in schoolwork, perform better academically, and have a more positive attitude toward school. Primary school students with specific learning difficulties have been reported to have lower self-efficacy beliefs than their peers.

Another perspective on self-evaluation and perception of difficulties can be explored through the concept of self-compassion. Neff defines self-compassion as a multifaceted construct that encompasses how individuals emotionally respond to suffering, cognitively understand their predicament, and pay attention to their suffering. A longitudinal study found that ninth-grade students with low self-esteem but high self-compassion exhibited better psychological health one year later compared to those with low self-compassion. Self-compassion has demonstrated its utility as a framework for interventions.

The aim of BEATLE is to provide understanding, inspiration, and tools for better learning in adolescents. This study aims to (1) analyze the effectiveness and feasibility of the BEATLE online rehabilitative course in three clinical groups (DLD, Dyslexia, and Mixed Specific Developmental Disorder) and (2) explore the potential differences in effectiveness among these diagnostic groups. For example, participants with dyslexia may report better and more lasting outcomes than participants with DLD or Mixed Specific Developmental Disorder, considering that the DCP includes several strategies for using digital tools such as dictation and text-to-speech, which can aid with primary difficulties related to reading and writing.

The study will employ a randomized controlled trial with a waitlist design. The objective is to assess potential changes in perceived self-efficacy, self-compassion, executive functioning, and attitudes toward learning as reported by participants, guardians (parents), and teachers. Additionally, this study aims to examine the correlation between the usage of the DCP and its effectiveness.

Participants will be recruited from 12-16-year-old patients referred to HUS Phoniatrics or HUS Pediatric Neurology. The target sample size is 52 participants per group (26 in the intervention group and 26 in the waitlist group), totaling 156 complete participants. Accounting for a conservative dropout rate of 50%, up to 312 participants may be required for recruitment. Another digital health program (DHP) on acquired brain injury patients in adults has reported a dropout rate of approximately 20%.

Recruitment will be conducted by neuropsychologists at respective clinics. After expressing willingness to participate, participants and their guardians will sign consent forms. Participants will then receive an envelope containing study materials and a consent form for their teacher to sign. Participation in the study does not supersede any other treatment.

Signed consent forms will be submitted to the research team, after which participants will be randomized into either the intervention group or the waitlist group. Randomization will be conducted in RedCap to minimize the risk of bias. Participants in the intervention group will receive an invitation to the DCP a few days after signing the agreement and completing the pre-intervention questionnaires. Participants in the waitlist group will first complete baseline questionnaires and will then wait 10 weeks before entering the cross-over phase and receiving access to the DCP.

ELIGIBILITY:
For inclusion, the International Classification of Diseases 10th edition (ICD-10; WHO, 2018) diagnostic criteria accompanied with Finnish Current Care Guidelines will be used as follows:

Developmental Language Disorder Verbal reasoning skills (Verbal Reasoning Index = VCI) 1.5 standard deviations lower than average (< 78 Index points) Intact non-verbal reasoning skills (Perceptual Reasoning Index = PRI) > 84 index points) Normal or fixed to normal hearing and vision Adequate skills in Finnish: Finnish either as a native language, major household language or adequate reported performance in Finnish school system.

Dyslexia Measured reading accuracy and comprehension two standard deviations (-2 standard deviations) lower than anticipated when the chronological age and IQ have been taken into account Normal of fixed to normal hearing and vision Adequate skills in Finnish: Finnish either as a native language, major household language or adequate reported performance in Finnish school system.

Mixed Developmental Disorder Wide developmental and learning difficulties (69 < PRI < 84, 69 < VCI < 84) Normal or fixed to normal hearing and vision Adequate skills in Finnish: Finnish either as a native language, major household language or adequate reported performance in Finnish school system.

Exclusion Criteria:

All exclusion criteria will be addressed individually. If a respondent fulfills one or more of the exclusion criteria, the respondent will be dropped out. Exclusion criteria are formed as follows:

Suspicion of mild intellectual disability Both verbal and non-verbal reasoning skills more than two standard deviations lower than average (VCI & PRI < 70) Weak (-2 Standard Deviations) performance on both subtests representing fluid intelligence (Wechsler's Intelligence Scale for Children IV (WISC-IV): Matrix reasoning and Picture concepts)

Diagnosis of Autism Spectrum Disorder

Untreated Attention-Deficit Hyperactivity Disorder

Unable to adequately use a a computer and/or a smartphone

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 312 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy Questionnaire for Children and Adolescents (SEQ-C) | Filled three to four times in different phases of the study. Both arms fill the measure before the intervention, after intervention and three months after the intervention. Waitlist- arm also fills the measure on the start of the waitlist period.
  A brief questionnaire assessing perceived academic, emotional and social self-efficacy. Scale scores will be calulated for academic (Min 8 - Max 40), emotional ( Min 7 - 35) and social self-efficacy (Min 8 - Max 40). A total self-efficacy score will also be calculated as a sum of abovementioned three scale scores (Min 23 - Max 115).
Sussex-Oxford Compassion Scale - Self (SOCS-S) | Filled three to four times in different phases of the study. Both arms fill the measure before the intervention, after intervention and three months after the intervention. Waitlist- arm also fills the measure on the start of the waitlist period.
  A brief questionnaire intended to measure perceived self-compassion. The measure consists of 20 items that are answered on 5-step likert scale. Five scale sum scores will be calculated from the measure: Recognition of suffering (Min 4 - Max 20), Understanding the universality of suffering (Min 4 - Max 20), Feeling sympathy for those who are suffering (Min 4 - Max 20), Tolerating the distress associated with the witnessing of suffering (Min 4 - Max 20) and Motivation to act to alleviate the suffering (Min 4 - Max 20). A total self-compassion score will also be calculated that is the sum of above mentioned five scale scores (Min 20 - Max 100).

SECONDARY OUTCOMES:
5-15 | Filled three to four times in different phases of the study. Both arms fill the measure before the intervention, after intervention and three months after the intervention. Waitlist- arm also fills the measure on the start of the waitlist period.
  5-15 is a questionnaire designed to assess perceived difficulties in children or adolescents. Parents and teachers of the participant will fill parts of this survey regarding executive functioning and learning. All items are answered on a three-step scale from 0 to 2.
  Following scale sum variables will be calculated:
  Reading, writing, calculating (13 items: MIN 0 - MAX 26), Learning and participation in learning (6 items: MIN 0 - MAX 12), Problem solving in learning situations (10 items: MIN 0 - MAX 20).
The Strengths and Difficulties Questionnaire (SDQ) | Filled three to four times in different phases of the study. Both arms fill the measure before the intervention, after intervention and three months after the intervention. Waitlist- arm also fills the measure on the start of the waitlist period.
  The Strengths and Difficulties Questionnaire is a brief behavioural screening questionnaire about 2-17 year olds. Parent and teacher of the participant is given SDQ to be filled in different timepoints of the study. SDQ consists of 25 symptom items that are answered on three-step scale from 0 to 2 and provide five scale sum scores to be calculated: Emotional difficulties scale (MIN 0 - MAX 10), Conduct difficulties scale (MIN 0 - MAX 10), Hyperactivity scale (MIN 0 - MAX 10), Peer difficulties scale (MIN 0 - MAX 10), Prosocial Scale (MIN 0 - MAX 10). A total difficulties score is also calculated by summing scores from all symptom scales except the prosocial scale (MIN 0 - MAX 40). Internalizing score ranges from 0 to 20 and is the sum of emotional and peer difficulties scales. The externalizing score ranges from 0 to 20 and is the sum of the conduct and hyperactivity scales.

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Pediatric Neurology, Helsinki University Hospital, Helsinki
  - Phoniatrics, Helsinki University Hospital, Helsinki

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are in favor of sharing anonymized individual participant data (IPD) collected in this study. However, the process for data sharing is still under review, and guidance is being sought on the permitted methods for making anonymized data available. Once the regulatory and institutional guidelines are clarified, a decision will be made regarding the extent and format of data sharing. If data sharing is approved, details on access procedures, including any necessary agreements or repositories used, will be provided in the study record.